CLINICAL TRIAL: NCT03449641
Title: PAP Therapy Compliance in Patients With Obesity Hypoventilation Syndrome
Brief Title: PAP Therapy in Patients With Obesity Hypoventilation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Principal Investigator, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSPAP1
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive airway pressure (PAP) treatment (Other): Positive airway pressure (PAP),which reverses upper airway obstruction, is effective in the majority of patients with stable obesity hypoventilation syndrome (OHS).
  Interventions: Device: Positive airway pressure (PAP)

INTERVENTIONS:
Device: Positive airway pressure (PAP) — Positive airway pressure (PAP) is a mode of respiratory ventilation used in the treatment of sleep apnea.

SUMMARY:
The role of different levels of compliance and long-term effects of positive airway pressure (PAP) therapy on gas exchange, sleepiness, quality of life, depression and death rate in patients with obesity hypoventilation syndrome (OHS).

DETAILED DESCRIPTION:
Various forms of positive airway pressure (PAP) therapy are effective in providing short and long-term benefits in these patients with or without obstructive sleep apnea (OSA). However, there are limited data concerning the impact of long-term effects of PAP therapy on survival and functional status in individuals with obesity hypoventilation syndrome (OHS) and OSA. Therefore we aimed to assess the role of different levels of compliance and long-term effects of PAP on gas exchange, sleepiness, quality of life, depression and death rate in patients with OHS, two year after PAP initiation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years
* Obesity hypoventilation syndrome diagnosis (OHS)
* clinically stable for at least 4 weeks prior to the enrolmenT
* above-elementary school education.

Exclusion Criteria:

* refusal to participate
* refusal of PAP therapy
* central sleep apnea syndromes
* restrictive ventilation syndromes
* severe congestive heart failure
* a history of life-threatening arrhythmias
* severe cardiomyopathy
* significant chronic kidney disease
* untreated hypothyroidism
* family or personal history of mental illness
* drug or alcohol abuse
* sedative use
* severe cognitive impairment
* concurrent oncological diseases
* history of narcolepsy or restless legs syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Effects of positive airway pressure (PAP) therapy on gas exchange | 2 years
  Effects of positive airway pressure (PAP) therapy on arterial blood gases measurements

SECONDARY OUTCOMES:
Effects of positive airway pressure (PAP) therapy on sleepiness | 2 years
  Effects of positive airway pressure (PAP) therapy on epwoth Sleepiness scale score
Effects of positive airway pressure (PAP) therapy on quality of life | 2 years
  Effects of positive airway pressure (PAP) therapy on Short Form -36 questionnaire
Effects of positive airway pressure (PAP) therapy on depression | 2 years
  Effects of positive airway pressure (PAP) therapy on Beck Depression Inventory questionnaire
Effects of positive airway pressure (PAP) therapy on death rate | 2 years
  Effects of positive airway pressure (PAP) therapy on number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Schiza, MD, PhD, Study Chair — University of Crete

REFERENCES:
- [Derived] Bouloukaki I, Mermigkis C, Michelakis S, Moniaki V, Mauroudi E, Tzanakis N, Schiza SE. The Association Between Adherence to Positive Airway Pressure Therapy and Long-Term Outcomes in Patients With Obesity Hypoventilation Syndrome: A Prospective Observational Study. J Clin Sleep Med. 2018 Sep 15;14(9):1539-1550. doi: 10.5664/jcsm.7332. PMID 30176976